CLINICAL TRIAL: NCT03679897
Title: 0.25% Levobupivacaine Versus 0.375% Ropivacaine: a Comparative Study in Ultrasound-Guided Infraclavicular Brachial Plexus Block
Brief Title: Comparison of 0.375% Ropivacaine and 0.25% Levobupivacaine for Infraclavicular Brachial Plexus Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, Clinical Instructor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-1117
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Regional Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine group (Experimental): BPB with 0.375% ropivacaine solution
  Interventions: Drug: Ropivacaine solution
- Levobupivacaine group (Active Comparator): BPB with 0.25% levobupivacaine solution
  Interventions: Drug: Levobupivacaine solution

INTERVENTIONS:
Drug: Ropivacaine solution — ultrasound-guided infraclavicular brachial plexus block with 0.375% ropivacaine solution
  Other Names: rop
  Arms: Ropivacaine group
Drug: Levobupivacaine solution — ultrasound-guided infraclavicular brachial plexus block with 0.25% levobupivacaine solution
  Other Names: levo
  Arms: Levobupivacaine group

SUMMARY:
Infraclavicular brachial plexus block has been used more frequently with the development of high-resolution ultrasound. Compared with peripheral nerve block using landmark technique or nerve stimulator technique, ultrasound-guided peripheral nerve block decreases the required dose of local anesthetics. As the dose of the drug used decreases, the systemic toxic effects of local anesthetics are reduced. However, the decreased dose of the drugs might have influence on the onset time of local anesthetics. Thus, the investigator aimed to evaluated the onset time of the two equipotent local anesthetics, 0.375% ropivacaine and 0.25% levobupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1-3
* Patients undergoing upper extremity surgery with infraclavicular brachial plexus block

Exclusion Criteria:

* Patients who do not agree to participate in clinical trial
* Patients presenting with neurological deficits of the upper arm, severe coagulopathy, chronic renal failure, cardiopulmonary compromise, cerebral vascular disease, hypersensitivity to hyaluronidase or local anesthetics or local infection at the site of the infraclavicular block, pregnancy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-08 (Actual)

PRIMARY OUTCOMES:
onset time of sensory block | up to 40 minutes
  sensory block of 4 nerves(radial, median, ulnar, musculocutaneous nerve) was assessed with pin-prick test every 5 minutes till 40 minutes from the completion of drug injection

SECONDARY OUTCOMES:
onset time of motor block | up to 40 minutes
  motor block of 4 nerves(radial, median, ulnar, musculocutaneous nerve) was assessed with movement of fingers and elbow every 5 minutes till 40 minutes from the completion of drug injection
duration of analgesia | 24 hours
  defined as time for first request by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Won Uk Koh, M.D., Ph.D., Principal Investigator — University of Ulsan, College of Medicine, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Lee S, Chin KJ, Kim JS, Kim H, Ro YJ, Koh WU. Comparison of the onset time between 0.375% ropivacaine and 0.25% levobupivacaine for ultrasound-guided infraclavicular brachial plexus block: a randomized-controlled trial. Sci Rep. 2021 Feb 25;11(1):4703. doi: 10.1038/s41598-021-84172-2. PMID 33633231